CLINICAL TRIAL: NCT02440139
Title: Computer-Aided System for the Improvement of Nodule Detection and Characterization in Thoracic CT Based on a Novel Vessel Suppressed CT Volume
Brief Title: Evaluation of Computer-Aided Lung Nodule Detection Software in Thoracic CT for Riverain Technologies LLC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Polytechnic Institute and State University (Other)
Collaborators: Riverain Technologies (Industry)
Responsible Party: Principal Investigator, ShihChung Ben Lo, Adjunct Professor, Virginia Polytechnic Institute and State University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 458420
Record Dates: First submitted 2015-04-15; First posted 2015-05-12 (Estimated); Results first posted 2021-10-04 (Actual); Last update posted 2021-11-04 (Actual); Status verified 2021-11

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm 1 (No Intervention): Participating radiologists will perform clinical reading on ~300 cases. They will mark all locations of concern (clinically actionable nodules) on conventional thoracic CT images. Computer will measure time, readers score regions according to action and suspiciousness.
- Arm 2 (Active Comparator): Participating radiologists will perform clinical reading on ~300 cases. They will mark all locations of concern (clinically actionable nodules) on thoracic CT images aided by ClearRead CT Insight software as the intervention. Computer will measure time, readers score regions according to action and suspiciousness.
  Interventions: Device: ClearRead CT Insight

INTERVENTIONS:
Device: ClearRead CT Insight — During the second reading session (concurrent read), the radiologist will be presented with a standard appearing CT with CADe marks placed and the vessel suppressed same slice with the vessel suppressed view as the intervention. The second image, vessel suppressed, will be grayed out until the radiologist move the mouse to the second panel. The radiologist will mark locations. These may or may not correspond to the locations of the CAD markers. As before, the radiologist will assign a level of suspicious to each mark and indicate the need, if any, of an additional diagnostic action (CT Follow-up, Contrast CT, PET-CT, or Biopsy).
  Arms: Arm 2

SUMMARY:
STUDY DESIGN:

This is a retrospective, multi-reader, multi-case, (MRMC) randomized reader study.

OBJECTIVE:

Primary: The primary objective of this clinical study is to prove that a user aided with ClearRead CT InSight (CRCTI) is superior to the unaided reader for detecting actionable lung nodules.

Secondary: The secondary objective of this clinical study is to prove that the reader's reading time is not significantly increased when aided with CRCTI.

NUMBER OF SUBJECTS:

Retrospective CT studies from approximately 300 patients will be included in the study. Approximately 100 true positive cases and 200 normal cases.

NUMBER OF READERS:

A reader study with at least ten (10) participating radiologists (US Board Certified) will be conducted.

PRIMARY ENDPOINTS:

Scores given by the radiologists with and without ClearRead CT Insight will be recorded and compared to the true status of the study-cases. The frequency of the scores for each method (Unaided, Aided) will be tabulated and LROC curves constructed along with sensitivity, specificity, PPV, NPV and clinical actions. Additionally, machine nodule detection rate and false positives per patient on normal cases will be measured.

PATIENT POPULATION :

The study will target approximately one hundred (100) patients whose CT nodules were shown to be cancer and two hundred (200) normal patients. The patient population will be consistent with the national lung cancer screening protocols.

DETAILED DESCRIPTION:
A reader study with at least ten (10) participating radiologists will be conducted. A localized receiver operating characteristic curve will be used to evaluate radiologists' diagnostic performance (in terms of the trade-off between the sensitivity and specificity when the decision criteria changes) in the detection of lung nodules on lung CTs with and without the usage of the ClearRead CT Insight (CRCTI) system. The time needed for the review and interpretation of each case will also be recorded.

An initial (baseline) interpretation will be made by each of the radiologists based on the Lung CT in its original form. At a minimum of one month later, each radiologists will again interpret the same images viewing the pair of CRCTI CT series: Two sets of CT images (standard with CADe marks and processed with vessel suppression will be presented on either one large monitor or two adjacent monitors.

During the baseline reading the radiologist will mark the location of the actionable nodules and assign a score. The radiologist will also indicate the recommended method of follow-up (Contrast CT, PET-CT, CT Follow-up, Biopsy).

During the second reading session (concurrent read), the radiologist will be presented with a standard appearing CT with computer-aided detection (CADe) marks placed and the vessel suppressed same slice with the vessel suppressed view (right image). The second image, vessel suppressed, will be grayed out until the radiologist move the mouse to the second panel. The radiologist will mark locations. These may or may not correspond to the locations of the CAD markers. As before, the radiologist will assign a level of suspicious to each mark and indicate the need, if any, of an additional diagnostic action (CT Follow-up, Contrast CT, PET-CT, or Biopsy).

Based on the levels of suspicion for each nodule and the associated likelihood ratings, LROC curves will be constructed for both the baseline and the concurrent reads and the significance of any difference will be calculated. The recommendations for further action (CT Follow-up, Contrast CT, PET-CT, or Biopsy) will be used to calculate sensitivity and specificity, PPV and NPV.

Number and types of cases:

Retrospective lung CT image series from approximately 300 patients will be included in the study. Approximately one hundred (100) of the patients will have pathology confirmed cancers and approximately two hundred (200) of the patients will be CTs associated with normal patients. Also included as nodule images are those where the actionable nodule was not acted on at that time, but was detected and acted on based on a subsequent CT. These are the prior images where the nodule can be identified and its location is the same as on the "current" image confirmed by the radiologist expert panel (using a majority of three as the decision criterion).

The selected sample, randomly selected from a larger pool of CT cases will be enriched in the following way:

1. Lung nodules (cancers in this study) will be tumor size T1a (20 mm or less). The proportion of nodules 20 mm or less may be increased since this is where the investigators expect the major impact of this software to be.
2. Non-Solid (ground glass) nodules will be added to the sample (based on availability) to determine the performance of the system on non-solid nodules. For this group, to have sufficient cases, the investigators may have to include benign (non-malignant) non-solid nodules.
3. In this project, the investigators will perform a Machine Test of the ClearRead CT Insight algorithm followed by a reader performance evaluation study. Riverain will provide a system configured with the operating point set to be used for the reader studies and a configuration for an "open" system to be used for machine testing and FROC generation.

Arm 1: a baseline read (no secondary content) and Arm 2: concurrent, CAD augmented read.

1. st Arm: Do baseline (measure time, readers score regions according to action and suspiciousness) - mark all locations of concern
2. nd Arm: Concurrent read (measure time, readers score regions according to action and suspiciousness) - mark all locations of concern

The primary study hypothesis is that the adjunctive use of ClearRead CT Insight is superior to use of standard lung CT images alone, as measured by the area under the LROC curve.

STATISTICAL ANALYSES Accuracy

To evaluate the hypothesis of superiority in terms of improvement in accuracy for ClearRead CT Insight vs. unaided, a mixed effects model (DBM) will be implemented (similar to the model outlined in Dorfman, Berbaum and Metz, 1997), where variance components will be included to account for reader, case, reader by case, reader by modality, case by modality and reader by case by modality. However, it is anticipated that the three-way interaction will be inestimable and will subsequently be dropped from the statistical model. Specifically, the hypothesis to test for superiority of ClearRead CT Insight vs. unaided is:

H0: AUCunaided - AUCClearRead CT Insight ≥ 0.0 vs. HA: AUCunaided - AUCClearRead CT Insight < 0

The AUC of the LROC is the primary endpoint to evaluate accuracy and the test of interest will be a two-sided 95% confidence interval on the effect of modality (i.e. ClearRead CT Insight minus unaided). Significance will be concluded if the upper bound of the two-sided 95% confidence interval does not include zero. If the null hypothesis (H0) is rejected, the alternative hypothesis (HA) is accepted and the superiority of using the ClearRead CT Insight system will be established.

Time

The second co-primary objective is to evaluate reduction in time spent per image for ClearRead CT Insight vs. unaided. Specifically, the hypothesis to test for superiority of ClearRead CT Insight vs. unaided is:

H0= Tunaided - TClearRead CT Insight ≤ 0 vs. HA= Tunaided - TClearRead CT Insight > 0

To evaluate the hypothesis of non-inferiority in terms of improved read time for ClearRead CT Insight vs. unaided, a mixed effects model will be implemented (similar to the model outlined in Dorfman, Berbaum and Metz, 1992), where variance components will be included to account for reader, case, reader by case, reader by modality, case by modality and reader by case by modality. However, it is anticipated that the three-way interaction will be inestimable and will subsequently be dropped from the statistical model.

The read times will be tested using a two-sided 95% confidence interval on the effect of modality (i.e. ClearRead minus unaided). Significance will be concluded if the upper bound of the two-sided 95% confidence interval does not include zero.

With either analysis, the use of the mixed model could be modified to employ a bootstrap sampling approach if the model assumptions of the DBM method have been violated. The upper 95 % confidence limit for the difference in the areas under the curves would be calculated using 10,000 bootstraps in the MultiReader MultiCase (MRMC) ROC method.

POWER AND SAMPLE SIZE

The power to detect differences in the AUC of the LROC curve for the proposed statistical analysis using the current design baseline, i.e. 300 cases, each corresponding image read by 10 readers, was assessed through a simulation study. Specifically, the model outlined above was used to simulate 500 datasets across a range of effect sizes, where power was defined as the proportion of datasets that yielded a significant p-value for testing the fixed effect of modality. The method of Dorfman, Berbaum and Metz, 1992 (DBM) was implemented utilizing statistical mixed model theory with jackknife estimates.

These simulations required assumptions regarding the magnitude of the variance components associated with the different random effects. As a pilot study to obtain estimates of variance components was not conducted, variance component estimates from Riverain study SoftView 510(k) (Record # BSSI-PR-09-00006) that uses a similar technology as the proposed ClearRead CT Insight device were used in all power simulations. Please note that the variance components were scaled by the total variance to represent the proportion of total variance explained by each component. All power estimates are dependent upon the appropriateness of the assumed variance components.

ELIGIBILITY:
Inclusion Criteria:

A thoracic CT case that is associated or with a feature of the following:

1. Asymptomatic patients age 55 - 77 with history of smoking
2. Primary Lung Cancer
3. Biopsy Proven (LuRADS 5) with radiology report
4. Screen detected event plus 1 prior CT. 2 year of prior CTs is preferred, if available.
5. <= 3mm slice spacing, no gaps
6. Use standard reconstruction kernels
7. Maximum of 5 nodules per image
8. Nodules must be 5-20mm in size
9. With or without contrast

Exclusion Criteria:

Thoracic CT cases that meet the following exclusion criteria will not be collected for use during clinical testing.

1. No Acute pneumothorax
2. Both lungs must be fully visible within the field of view
3. Apices cannot be cropped
4. No excessive motion artifacts
5. Symptomatic patients with co-morbidities

Ages: 55 Years to 77 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2015-04; Primary Completion 2017-09 (Actual); Study Completion 2018-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew T Freedman, M.D., Study Director — Virginia Polytechnic Institute and State University
Locations (1):
- Arlington Innovation Center: Health Resaerch, Arlington, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Beyer F, Zierott L, Fallenberg EM, Juergens KU, Stoeckel J, Heindel W, Wormanns D. Comparison of sensitivity and reading time for the use of computer-aided detection (CAD) of pulmonary nodules at MDCT as concurrent or second reader. Eur Radiol. 2007 Nov;17(11):2941-7. doi: 10.1007/s00330-007-0667-1. Epub 2007 May 22. PMID 17929026
- [Background] Dorfman DD, Berbaum KS, Metz CE. Receiver operating characteristic rating analysis. Generalization to the population of readers and patients with the jackknife method. Invest Radiol. 1992 Sep;27(9):723-31. No abstract available. PMID 1399456
- [Background] Foti G, Faccioli N, D'Onofrio M, Contro A, Milazzo T, Pozzi Mucelli R. Evaluation of a method of computer-aided detection (CAD) of pulmonary nodules with computed tomography. Radiol Med. 2010 Sep;115(6):950-61. doi: 10.1007/s11547-010-0556-6. Epub 2010 Jun 23. English, Italian. PMID 20574707
- [Background] Matsumoto S, Ohno Y, Aoki T, Yamagata H, Nogami M, Matsumoto K, Yamashita Y, Sugimura K. Computer-aided detection of lung nodules on multidetector CT in concurrent-reader and second-reader modes: a comparative study. Eur J Radiol. 2013 Aug;82(8):1332-7. doi: 10.1016/j.ejrad.2013.02.005. Epub 2013 Mar 6. PMID 23480965
- [Background] Obuchowski NA. New methodological tools for multiple-reader ROC studies. Radiology. 2007 Apr;243(1):10-2. doi: 10.1148/radiol.2432060387. No abstract available. PMID 17392244
- [Background] Obuchowski NA, McClish DK. Sample size determination for diagnostic accuracy studies involving binormal ROC curve indices. Stat Med. 1997 Jul 15;16(13):1529-42. doi: 10.1002/(sici)1097-0258(19970715)16:133.0.co;2-h. PMID 9249923

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 12 radiologists were invited to participate in a two-arms reader study.
Units Other Than Participants: CT cases
Groups:
- Arm 1: Participating radiologists performed clinical reading on 328 cases. They marked all locations of concern (clinically actionable nodules) on conventional thoracic CT images. Computer measured time, readers score regions according to action and suspiciousness.
Period: Overall Study
Arm/Group | Arm 1
Started (June 2015) | 12; 324 CT cases (12 radiologists read 324 CT cases)
Completed (August 2016) | 12; 324 CT cases (12 radiologists read 324 CT cases)
Not Completed | 0; 0 CT cases

BASELINE CHARACTERISTICS:
Population: 12 US board-certified radiologists were invited to participate in the study. They were 8 males and 4 females.
Groups:
- Arm 1: Baseline Study: 12 participating radiologists performed clinical reading on 324 cases. They marked all locations of concern (clinically actionable nodules) on conventional thoracic CT images. Computer measured time, readers score regions according to action and suspiciousness.
Arm/Group | Arm 1: Baseline Study
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 12
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 8
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: Comparing the Detection Accuracy, Sensitivity, and Specificity of Clinically Actionable Lung Nodules
Description: The detection rates in accuracy, sensitivity, and specificity on clinically actionable lung nodules were computed and compared for Aim 1 (baseline) and Arm 2 (study participants were aided with ClearRead CT software) studies.
Time Frame: 4 months
Population: Of the study chest CT cases, some contained cancers and/or clinically actionable benign nodules. They were considered targets in the study. The remaining study cases had no cancer nor clinically actionable nodules which served as true-negative for the study.
Measure: Count of Units; unit: CT-case | nodule
Units Other Than Participants: CT-case | nodule
Groups:
- Arm 1: Participating radiologists performed a clinical reading on the study cases. They marked all locations of concern (clinically actionable nodules) on conventional thoracic CT images. Computer measured time, readers score regions according to action and suspiciousness.
- Arm 2: Participating radiologists performed clinical reading on the study cases. They marked all locations of concern (clinically actionable nodules) on thoracic CT images aided by ClearRead CT Insight software as the intervention. Computer measured time, readers score regions according to action and suspiciousness.
  ClearRead CT Insight: During the second reading session (concurrent read), the radiologist was presented with a standard appearing CT with CADe marks placed and the vessel suppressed images with the vessel suppressed view as the intervention. The second image, vessel suppressed, was not shown until the radiologist move the mouse to the second panel. The radiologist will mark locations. These may or may not correspond to the locations of the CAD markers. As before, the radiologist then assigned a level of suspicious to each mark and indicate the need, if any, of an additional diagnostic action (CT Follow-up, Contrast CT, PET-CT, or Biopsy).
Arm/Group | Arm 1 | Arm 2
Number analyzed (Participants) | 12 | 12
Number analyzed (CT-case | nodule) | 4728 | 4728
CT-case | nodule
  Detection Accuracy | 3612 | 3735
  Detection Sensitivity: number analyzed (CT-case | nodule) | 2136 | 2136
  Detection Sensitivity | 1283 | 1548
  Detection Specificity: number analyzed (CT-case | nodule) | 2592 | 2592
  Detection Specificity | 2329 | 2187
Statistical Analysis 1: Comparison: Arm 1 vs Arm 2; Test type: Superiority; p < 0.05, Mixed Models Analysis; difference in sensitivity = -0.124, 95% CI 2-sided [-0.186 to -0.062], Standard Deviation 0.034

2. Primary Outcome: Comparing LROC Curve in the Detection of Clinically Actionable Lung Nodules Among Normal
Description: The areas under location-specific Receiver Operating Characteristic (LROC) curves were computed and compared for Aim 1 (baseline) and Aim 2 (study participants were aided with ClearRead CT software).
Time Frame: 4 months
Measure: Geometric Mean (95% Confidence Interval); unit: Probability
Units Other Than Participants: CT case
Groups:
- Arm 1: Participating radiologists performed a clinical reading on the study cases. They will mark all locations of concern (clinically actionable nodules) on conventional thoracic CT images. Computer measured time, readers score regions according to action and suspiciousness.
- Arm 2: Participating radiologists performed a clinical reading on the study cases. They marked all locations of concern (clinically actionable nodules) on thoracic CT images aided by ClearRead CT Insight software as the intervention. Computer measured time, readers score regions according to action and suspiciousness.
  ClearRead CT Insight: During the second reading session (concurrent read), the radiologist was presented with a standard appearing CT with CADe marks placed and the vessel suppressed the same slice with the vessel suppressed view as the intervention. The second image, vessel suppressed, was not shown until the radiologist moves the mouse to the second panel. The radiologist will mark locations. These may or may not correspond to the locations of the CAD markers. As before, the radiologist then assigned a level of suspicion to each mark and indicate the need, if any, for an additional diagnostic action (CT Follow-up, Contrast CT, PET-CT, or Biopsy).
Arm/Group | Arm 1 | Arm 2
Number analyzed (Participants) | 12 | 12
Number analyzed (CT case) | 3888 | 3888
Probability | 0.633 [0.594 to 0.672] | 0.773 [0.734 to 0.812]
Statistical Analysis 1: Comparison: Arm 1 vs Arm 2; For each study arm, the difference in the least-squares means of the two arms was estimated. A two-sided 95% confidence interval on this difference in study arms (i.e. unaided minus aided by the software) was used to test the hypothesis that the difference in the area under the LROC curve (AUC). The superiority of ClearRead CT will be concluded if the upper bound of the two-sided 95% confidence interval on the difference is less than zero; Test type: Superiority; p < 0.05, ANOVA; Difference in LROC curves = -0.14, 95% CI 2-sided [-0.209 to -0.071], Standard Deviation 0.039

3. Secondary Outcome: Average Reading Time Per Case
Description: The average reading times per reader per case were computed and comapred in both Aim 1 and Arm 2 (study participants were aided with ClearRead CT software) studies.
Time Frame: 4 months
Measure: Mean (95% Confidence Interval); unit: Second
Units Other Than Participants: CT case
Arm/Group | Arm 1 | Arm 2
Number analyzed (Participants) | 12 | 12
Number analyzed (CT case) | 3888 | 3888
Second | 98.0 [88.0 to 108.0] | 132.3 [122.3 to 142.3]

ADVERSE EVENTS:
Time Frame: 4 months
Description: No adverse event occurred.
Groups:
- Arm 1: 12 Participating radiologists performed a clinical reading on 324 cases. They marked all locations of concern (clinically actionable nodules) on conventional thoracic CT images. Computer measured time, readers score, and regions according to action and suspiciousness.
- Arm 2: 12 Participating radiologists performed clinical reading on 324 cases. They marked all locations of concern (clinically actionable nodules) on thoracic CT images aided by ClearRead CT Insight software as the intervention. Computer measured time, readers score, and regions according to action and suspiciousness.
  ClearRead CT Insight: During the second reading session (concurrent read), the radiologist was presented with a standard appearing CT with CADe marks placed and the vessel suppressed the same slice with the vessel suppressed view as the intervention. The second image, vessel suppressed, was not shown until the radiologist moved the mouse to the second panel. The radiologist again marked locations. These may or may not correspond to the locations of the CAD markers. As before, the radiologist then assigned a level of suspicious to each mark and indicate the need, if any, of an additional diagnostic action (CT Follow-up, Contrast CT, PET-CT, or Biopsy).
Arm/Group | Arm 1 | Arm 2
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 0/12 | 0/12

LIMITATIONS AND CAVEATS:
This study only used a relatively low number of thoracic CT cases read by 12 radiologists. The study cases were mainly collected from the National Lung Screen Trial (NLST) lung cancer screening program. In addition, the study suffered from readers' lack of learning time of using the AI software.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-08-24): https://cdn.clinicaltrials.gov/large-docs/39/NCT02440139/Prot_SAP_000.pdf